CLINICAL TRIAL: NCT05546814
Title: Impact of Dietary Sodium Supplementation on Growth & Intestinal Microbiome in Preterm Infants
Brief Title: Impact of Dietary Sodium Supplementation on Growth & Intestinal Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Jeffrey Segar, Principal Investigator, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRBNet 1846631
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-04

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Two cohorts; experimental and control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Sodium algorithm (Experimental): Starting at 2 weeks of age, the sodium algorithm group will be started based on their sodium levels. This will be adjusted weekly based on weight gain and sodium levels.
  Interventions: Procedure: Sodium algorithm
- Control (No Intervention): Subjects will be cared for by current protocols

INTERVENTIONS:
Procedure: Sodium algorithm — Infants will receive sodium and follow a sodium supplementation schedule or algorithm. This means that based on the sodium levels collected from the samples (stool and urine) they will receive an increase or maintain the same amount to help
  Arms: Sodium algorithm

SUMMARY:
The purpose of this project is to determine the direct impact of sodium supplementation in preterm infants and to see the overall improvement of their growth and health status.

from this study will help us develop a better treatment for in the future.

DETAILED DESCRIPTION:
Premature infants are at an increased risk of postnatal growth failure and as well as developing short or long-term impaired neurodevelopment and cardio metabolic health.

For many years, it has been recognized that ideal growth is attainable with sufficient sodium intake and a positive sodium balance. The results of this study could have a significant impact on the care of preterm infants.

Infants will be randomized into one of two groups. One group will receive sodium supplementation as guided by a urine sodium concentration algorithm, one group will be managed by current standards. Randomization will occur at 2 weeks of postnatal age

Standard of care group Care for the participant will remain the same as if they were not in the study. Nutritional information, including sodium intake will be collected on three separate days weekly for 8 weeks. Stool samples will be collected for determining intestinal microbiome at 2 weeks, 5 weeks, 8 weeks and the day they are discharged from the hospital.

The study team will also collect detailed health information from participants hospital stay from the medical chart. Which will include gestational age, birth weight, sex, race ,ethnicity, mode of delivery and exposure to any steroids, antibiotics and clinical diagnoses.

Sodium supplementation group:

Participants will receive sodium supplementation per the urine sodium concentration algorithm. Urine sodium will be determined weekly, and if urine sodium concentration is below set value, dietary sodium supplementation is provided.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight >500 grams and
* Gestational age at least 25 0/7weeks but less than 30 weeks.
* <14 days of age at time of randomization

Exclusion Criteria:

* Non-English speaking parents
* Major congenital anomalies
* grade underlying renal dysfunction (serum creatinine > 1.0 mg/dL or increase of >0.3 mg/DL between any two consecutive measurements)
* use of diuretics at the time initiation of intervention (approximately 14 days of age) But this is not completely an exclusion-the research can wait 2 days and at the time of 2 week time period of the study we can re check their levels
* any structural genitourinary criteria.

Ages: 25 Weeks to 30 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

PRIMARY OUTCOMES:
Preterm infant weight gain | 8 weeks
  To determine the relationship among sodium intake, bodily growth and the gut in preterm infants

SECONDARY OUTCOMES:
Microbiome | 8 weeks
  Microbiome diversity according to study group

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Segar, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No